CLINICAL TRIAL: NCT07322289
Title: Evaluating the Use of Antibiotic-Coated Braided Sutures in Debridement, Antibiotic, and Implant Retention (DAIR) Procedures
Brief Title: Antibiotic-coated Braided Suture Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Colin A. McNamara, Assistant Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20250980
Record Dates: First submitted 2026-01-05; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Prosthetic Joint Infection; Debridement With Prosthesis Retention; Prosthetic Joint Infections of Hip; Prosthetic Joint Infections of Knee; Suture
Keywords: prosthetic joint infection; debridement, antibiotics, implant retention; antibiotic coated braided sutures; monofilament suture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Triclosan-Braided Suture Group (Experimental): Patients randomized to this arm will receive triclosan-coated braided sutures for closure of the fascia. Following incision and full debridement and irrigation, the fascia will be closed with this suture. Suturing of the fascia typically takes ~10 minutes. As this suture is absorbable, it does not have to be removed. The superficial layers of the skin will be closed with nylon suture.
  Interventions: Device: VICRYL™ Plus (Coated VICRYL™ Plus Antibacterial)
- Monofilament Suture Group (Active Comparator): Patients randomized to this arm will receive monofilament sutures for closure of the fascia. Following incision and full debridement and irrigation, the fascia will be closed with this suture. Suturing of the fascia typically takes ~10 minutes. As this suture is absorbable, it does not have to be removed. The superficial layers of the skin will be closed with nylon suture.
  Interventions: Device: Polydioxanone (PDS™ II ) Sterile Synthetic Absorbable Surgical Suture-Monofilament

INTERVENTIONS:
Device: VICRYL™ Plus (Coated VICRYL™ Plus Antibacterial) — Synthetic, absorbable, braided suture coated with triclosan for antimicrobial protection. Used for fascial and skin closure. Offers high tensile strength and knot security
  Arms: Triclosan-Braided Suture Group
Device: Polydioxanone (PDS™ II ) Sterile Synthetic Absorbable Surgical Suture-Monofilament — Absorbable, non-braided suture. Used for fascial and skin closure.
  Arms: Monofilament Suture Group

SUMMARY:
The purpose of this study is to evaluate whether the use of antibiotic-coated (triclosan) braided sutures is non-inferior or potentially superior to standard monofilament sutures in patients with prosthetic joint infections (PJIs) managed with the DAIR protocol. Several studies in various surgical specialties have demonstrated the effectiveness and non-inferiority of triclosan-coated braided sutures in infected surgical cases, and the study intends to transpose this idea to the management of prosthetic joint infections. Monofilament sutures are the present standard of care in any infected joint case due their lower surface area for bacterial harborization, though surgeons sacrifice mechanical integrity and comfortability with the closure in the process. By demonstrating the safety of antibiotic -coated braided sutures, surgeons will no longer have to make this compromise.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Willing and able to provide informed consent
* Primary Total Hip Arthroplasty or Total Knee Arthroplasty with Prosthetic Joint Infection Musculoskeletal Infection Society (MSIS) criteria
* Prosthetic Joint Infection Treated with Debridement, Antibiotics, Implant Retention

Acute Prosthetic Joint Infection: <4 weeks since it was suspected/diagnosed

Exclusion Criteria:

* Staphylococcus aureus bacteremia
* Mycobacterial, fungal, or parasitic infection
* Concurrent infection needing prolonged Intravenous therapy
* Septic shock/systemic illness needing IV therapy
* Patients with severe immunosuppression (ex: chemotherapy,

neutropenia, HIV, steroid use

* Allergy to Triclosan
* Pregnancy
* Prisoners

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with treatment failure at 90 days | 90 days post treatment
  Treatment failure is defined by Musculoskeletal Infection Society Criteria for prosthetic joint infection, including persistent wound drainage, sinus tract formation, positive cultures, or need for surgical revision.The proportion will be calculated as the number of patients meeting any MSIS treatment-failure criterion divided by the total number of patients evaluated. Assessment will be based on clinical evaluation and microbiological data collected at 90 days post-treatment.

SECONDARY OUTCOMES:
Net Cost Comparison of Triclosan-Coated Braided vs. Monofilament Sutures (USD per patient) | Within 90 days of surgery
  A cost analysis will be conducted to compare the net expenses associated with the use of triclosan-coated braided absorbable sutures versus monofilament absorbable sutures for fascial and skin closure. The analysis will include direct material costs, operative time, and any postoperative complications requiring additional interventions.
Incidence of Wound Dehiscence | Up to 90 days post-operative
  Medical records will be reviewed for any documented wound dehiscence following surgery
Incidence of Superficial Site Infection | Up to 90 days post-operative
  Medical records will be reviewed for any documented superficial surgical site infection
Incidence of Seroma Formation | Up to 90 days post-operative
  Medical records will be reviewed for any documented seroma formation following surgery
Incidence of Delayed Wound Healing | Up to 90 days post-operative
  Medical records will be reviewed for any documented delayed wound healing

CONTACTS AND LOCATIONS:
Overall Officials: Colin McNamara, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Health System, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No